CLINICAL TRIAL: NCT01044654
Title: A Phase 1 Dose Escalation, Single Dose Study of Autologous T-Cells Genetically Modified at the CCR5 Gene by Zinc Finger Nucleases SB-278 in HIV-Infected Patients Who Have Exhibited Suboptimal CD4+ T-Cell Gains During Long-Term Antiretroviral Therapy
Brief Title: Phase 1 Dose Escalation Study of Autologous T-cells Genetically Modified at the CCR5 Gene by Zinc Finger Nucleases in HIV-Infected Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sangamo Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SB-728-0902
Record Dates: First submitted 2010-01-06; First posted 2010-01-08 (Estimated); Last update posted 2015-03-13 (Estimated); Status verified 2015-03

CONDITIONS: HIV Infection; HIV Infections
Keywords: HIV; Treatment Experienced
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort 1 (Experimental): 3 Subjects will receive a single infusion of 0.5-1.0 x 1010 SB-728-T
  Interventions: Genetic: SB-728-T
- Cohort 2 (Experimental): 3 Subjects will receive a single infusion of 2.0 x 1010 SB-728-T
  Interventions: Genetic: SB-728-T
- Cohort 3 (Experimental): 3 Subjects will receive a single infusion of 3.0 x 1010 SB-728-T
  Interventions: Genetic: SB-728-T
- Cohort 4 (Experimental): Up to 4 HAART failure subjects will receive a single intravenous infusion of 0.5 to 3.0 x 1010 SB-728-T
  Interventions: Genetic: SB-728-T
- Cohort 5 (Experimental): Up to 20 subjects with heterozygote CCR5 delta-32 mutation will receive a single intravenous infusion of 0.5 to 3.0 x 1010 SB-728-T.
  Cohort 5 subjects will undergo a structured treatment interruption 2 months following infusion in which their anti-retroviral therapy will be discontinued for 16 weeks. HAART will be reinstituted in subjects whose CD4+ cell counts drop to <350 cells/mm3 and/or whose HIV-RNA increases to >100,000 on three consecutive weekly measurements.
  At the end of the STI, subjects with a sustained detectable viral load will be reinstituted on HAART. Subjects with HIV RNA levels below the limit of detection will remain off HAART. Subjects with an undetectable viral load will remain off HAART until HIV RNA levels are detectable or their CD4 count drops below 350 cell/mm3 on three consecutive weekly measurements.
  Interventions: Genetic: SB-728-T

INTERVENTIONS:
Genetic: SB-728-T — Each infusion will be 5-30 billion ZFN modified CD4+ T-cells

SUMMARY:
This research study is being carried out to study a new way to possibly treat HIV. This agent is called a "Zinc Finger Nuclease" or ZFN for short. ZFNs are proteins that can delete another protein named CCR5. This CCR5 protein is required for certain types of HIV (CCR5 tropic) to enter into and infect your T-cells. T cells are one of the white blood cells used by the body to fight HIV. The most important of these are called "CD4 T-cells."

Some People are born without CCR5 on their T-cells. These people remain healthy and are resistant to infection with HIV. Other people have a low number of CCR5 on their T-cells, and their HIV disease is less severe and is slower to cause disease (AIDS).

Even with no detectable levels of HIV in the blood, HIV remains in some tissues in the body, primarily the gut tissue. HIV infects the CD4+ T-cells including in the blood and gut. The new treatment to be studied will involve removing white blood cell from the blood that contains CD4+ T-cells. The extracted CD4+ T-cells are then genetically modified by the ZFNs to be resistant to infection by HIV by removing the CCR5 gene from the surface of the CD4+ T cell where HIV enters the cell. Additional genetically modified cells are manufactured and then re-infused back into you. Researchers hope that these genetically modified cells will be resistant to infection by HIV and will be able to reproduce additional resistant CD4+ T-cells in your body.

Laboratory studies have shown that when CD4+ T-cells are modified with ZFNs, HIV is prevented from killing the CD4+ T-cells. On the basis of these laboratory results, thre is the potential that ZFNs may work in humans infected with HIV and improve their immune system by allowing their CD4+ T-cells to survive longer.

The purpose of this research study is to find out whether "zinc finger" modified CD4+ T-cells are safe to give to humans and find how "zinc finger" modified T-cell affects HIV.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV infection prior to study entry
* Must be willing to comply with study-mandated evaluations; including not changing their antiretroviral regimen (unless medically indicated) during the study period.

Cohort 1, 2 and 3 (Enrollment Completed)

Cohort 5:

* Must have received HAART therapy, and had undetectable viral loads for at least 1 year.
* HIV-1 RNA < 50 copies/mL obtained within 60 days prior to study entry performed with an ultrasensitive HIV-1 PCR assay.
* CD4+ T cell count >500 cells/mm3
* Heterozygous for the CCR5 delta-32 mutation
* On stable antiretroviral medication (no changes to treatment within 4 weeks of screening and willing to discontinue current antiretroviral therapy during the structured therapy interruption

Cohort 4

* On stable antiretroviral medication (no changes to treatment within 4 weeks of screening and willing to continue on current antiretroviral therapy through week 8 after infusion
* CD4+ T cell count >350 cells/mm3.
* HIV-1 >1,000 copies/mL at screen and not responding to current antiviral therapy (i.e. HIV-RNA plasma levels > 1000 copies/ml after at least 12 weeks of stable, unchanged ARV therapy).

Exclusion Criteria:

* Acute or chronic hepatitis B or hepatitis C infection
* Active or recent (in prior 6 months) AIDS defining complication.
* Any cancer or malignancy within the past 5 years, with the exception of successfully treated basal cell or squamous cell carcinoma of the skin or low grade (0 or 1) anal or cervical dysplasia.
* Current diagnosis of NYHA grade 3 or 4 CHF, uncontrolled angina or uncontrolled arrhythmias.
* History or any features on physical examination indicative of a bleeding diathesis.
* Previous treatment with any HIV experimental vaccine within 6 months prior to screening, or any previous gene therapy using an integrating vector.
* Use of chronic corticosteroids, hydroxyurea, or immunomodulating agents (e.g., interleukin-2, interferon-alpha or gamma, granulocyte colony stimulating factors, etc.) within 30 days prior to enrollment
* Breast-feeding, pregnant or unwilling to use acceptable methods of birth control for 6 months following the last infusion of SB-728-T cells.
* warfarin or any other medication that is likely to affect platelet function or other aspects of blood coagulation during the 2 week period prior to leukapheresis.
* Active drug or alcohol use or dependence
* Serious illness requiring systemic treatment and/or hospitalization within 30 days prior to study entry.
* Recent vaccination or intercurrent illness (within 5 weeks prior to infusion)
* Have an allergy or hypersensitivity to study product excipients (human serum albumin, DMSO and Dextran 40).
* Subjects who are currently taking maraviroc or have received maraviroc within 6 months prior to screening.

Cohort 4 only:

* HIV-1 RNA >1,000 copies/mL at screen and not responding to current antiviral therapy
* CD4+ T cell count >350 cells/mm3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Safety - Treatment related adverse events | 12 months after the first infusion

SECONDARY OUTCOMES:
Evaluate the long-term persistence and activity of CCR5 ZFN-modified autologous T-Cells | 12 months after the first infusion

CONTACTS AND LOCATIONS:
Overall Officials: Winson Tang, M.D., Study Director — Sangamo Therapeutics
Locations (9):
- United States (9):
  - UCLA Center for AIDS Research and Education, Los Angeles, California
  - Orange Coast Medical Group, Newport Beach, California
  - Quest Clinical Research, San Francisco, California
  - Circle CARE Center, LLC, Norwalk, Connecticut
  - Orlando Immunology Center, Orlando, Florida
  - Central West Clinical Research, Inc., St Louis, Missouri
  - Southwest CARE Center, Santa Fe, New Mexico
  - Ricky K Hsu, MD, PC, New York, New York
  - Gordon Crofoot, MD, PA, Houston, Texas